CLINICAL TRIAL: NCT02310646
Title: A Clinical Trial Gathering Insight of Patient Reported Factors That Influence Preference Following Once Daily Topical Treatment With LEO 90100 Aerosol Foam and Daivobet® Gel in Subjects With Psoriasis Vulgaris
Brief Title: Patient Insights Following Use of LEO 90100 Aerosol Foam and Daivobet® Gel in Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LP0053-1030
Record Dates: First submitted 2014-11-28; First posted 2014-12-08 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group 1 (Active Comparator): Day 1 to 7: LEO 90100 aerosol foam Day 8 to 14: Daivobet® gel
  Interventions: Drug: LEO 90100 Aerosol Foam; Drug: Daivobet® gel
- Treatment group 2 (Active Comparator): Day 1 to 7: Daivobet® gel Day 8 to 14: LEO 90100 aerosol foam
  Interventions: Drug: LEO 90100 Aerosol Foam; Drug: Daivobet® gel

INTERVENTIONS:
Drug: LEO 90100 Aerosol Foam — Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Aerosol Foam 60 g per can, applied once daily for one week
Drug: Daivobet® gel — Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Gel 60 g per bottle, applied once daily for one week.

SUMMARY:
To gather insight on how product attributes affect usability by investigating the factors that are thought to influence patient preference to topical anti-psoriatic treatments.

DETAILED DESCRIPTION:
An international, multi-centre, prospective, open-label, randomised, 2-arm, cross-over study with 14-days once daily treatment in subjects with psoriasis vulgaris. To gather insight on how product attributes affect usability by investigating the factors that are thought to influence patient preference to topical anti-psoriatic treatments.

ELIGIBILITY:
Inclusion:

1. At Day 1 (Visit 1), a clinical diagnosis of psoriasis vulgaris of at least 6 months duration involving the trunk and/or limbs amenable to treatment with a maximum of 60 g of study medication per week
2. Psoriasis vulgaris on the trunk and/or limbs (excluding psoriasis on the genitals and skin folds) involving 2-30% of the Body Surface Area (BSA) at Day 1 (Visit 1)
3. A Physician's Global Assessment of disease severity (PGA) of at least mild on trunk and/or limbs at Day 1 (Visit 1)
4. A modified PASI (m-PASI) score of at least 2 on the trunk and/or limbs at Day 1 (Visit 1)

Exclusion:

1. Topical anti-psoriatic treatment on the trunk and limbs within 2 weeks prior to randomisation.
2. Any previous topical treatment with calcipotriol plus betamethasone gel (Daivobet® gel or Xamiol® gel).
3. Psoralen combined with Ultraviolet A (PUVA) therapy within 4 weeks prior to randomisation.
4. Ultraviolet B (UVB) therapy within 2 weeks prior to randomisation.
5. Planned excessive exposure of area(s) to be treated with study medication to either natural or artificial sunlight (including tanning booths, sun lamps etc.) during the trial.
6. Subjects who have received treatment with any non-marketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to randomisation.
7. Previously randomised into a clinical trial involving LEO 90100.
8. Current participation in any other interventional clinical trial.
9. Previously randomised into this trial.
10. Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
11. Subjects with any of the following conditions present on the treatment area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ulcers and wounds.
12. Other inflammatory skin disorders (e.g. seborrhoeic dermatitis or contact dermatitis) on the treatment area that may confound the evaluation of psoriasis.
13. Known or suspected disorders of calcium metabolism associated with hypercalcaemia.
14. Known or suspected severe renal insufficiency or severe hepatic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Papp, MD phD, Principal Investigator — K. Papp Clinical Research INC.
Locations (1):
- K.Papp Clinical Research Inc., Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 219 subjects from Canada (8 sites) and Germany (7 sites) were enrolled into the trial. First Subject First Visit:10-Feb-2015 and Last Subject Last Visit: 03-Aug-2015 (last visit, including follow-up). 6 enrolled subjects were not randomised.
Pre-assignment Details: Screening assessments were performed at the Screening Visit which could occur up to 28 days prior to Baseline (Day 1; Visit 1). A washout period of up to 4 weeks was to be completed if the subject was treated or had recently been treated with anti-psoriatic treatments or other relevant medication, as defined by the exclusion criteria.
Groups:
- Foam - Gel: Day 1 to 7: LEO 90100 aerosol foam Day 8 to 14: Daivobet® gel
  LEO 90100 Aerosol Foam: Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Aerosol Foam 60 g per can, applied once daily for one week
  Daivobet® gel: Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Gel 60 g per bottle, applied once daily for one week.
- Gel - Foam: Day 1 to 7: Daivobet® gel Day 8 to 14: LEO 90100 aerosol foam
  LEO 90100 Aerosol Foam: Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Aerosol Foam 60 g per can, applied once daily for one week
  Daivobet® gel: Calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) Gel 60 g per bottle, applied once daily for one week.
Period: First Intervention (Day 1 - Day 7)
Arm/Group | Foam - Gel | Gel - Foam
Started | 109 | 104
Completed | 107 | 104
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention (Day 8 - Day 14)
Arm/Group | Foam - Gel | Gel - Foam
Started | 107 | 104
Completed | 107 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the foam-gel group discontinued from the trial prior to the Week 1 visit and did not complete any on-treatment questionnaires. This subject was excluded from the full analysis set which hence comprised 212 subjects: 108 subjects in the foam-gel group and 104 subjects in the gel-foam group.
Groups:
- Foam - Gel: Day 1 to 7: LEO 90100 aerosol foam Day 8 to 14: Daivobet® gel
- Gel - Foam: Day 1 to 7: Daivobet® gel Day 8 to 14: LEO 90100 aerosol foam
- Total: Total of all reporting groups
Arm/Group | Foam - Gel | Gel - Foam | Total
Number analyzed (Participants) | 108 | 104 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 81 | 162
  >=65 years | 27 | 23 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.0) | 51.6 (14.2) | 51.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 34 | 79
  Male | 63 | 70 | 133

OUTCOME MEASURES:

1. Primary Outcome: Overall Treatment Preference by Subject's Preference Assessment (SPA) at Week 2 and Association With Baseline Characteristics
Description: The SPA questionnaire was completed at Week 2 and consisted of 2 parts:
  (i) the subject indicated if they preferred LEO 90100 foam or Daivobet® gel based on their experience using these products for 1 week each during the 2-weeks treatment period; (ii) the subject indicated how much each of the 22 items under the application, formulation, and container domains contributed to their overall decision of which product they preferred. This part of the SPA tool used a 4-point scale ranging from 'very important factor' to 'not at all important factor'.
  The statistical significance of each of the following 7 baseline characteristics (gender, age, disease severity, distribution, plaque size, skin thickness, onset) was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors.
  Results of multiple regression analyses are provided in the Clinical Study Report which can be found on the LEO Pharma website.
Time Frame: 2 weeks
Measure: Number; unit: percentage of subjects
Groups:
- All Randomised Subjects: All randomised subjects (foam - gel and gel - foam)
Arm/Group | All Randomised Subjects | Foam - Gel | Gel - Foam
Number analyzed (Participants) | 212 | 108 | 104
percentage of subjects
  Overall, I preferred the aerosol foam | 49.5 | 52.9 | 46.2
  Overall, I preferred the gel in a bottle | 50.5 | 47.1 | 53.8
Statistical Analysis 1: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: gender (male, female); Test type: Superiority or Other; p = 0.2, Regression, Logistic — Treatment sequence effect: p=0.28; gender effect: p=0.20; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and gender as factors
Statistical Analysis 2: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: age (18-39 years, 40-59 years, ≥60 years); Test type: Superiority or Other; p = 0.001, Regression, Logistic — Treatment sequence effect: p=0.34; age effect: p=0.001; threshold for statistical significance: p<0.05; 2-factor logistic regression with age and treatment sequence as factors
Statistical Analysis 3: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: Baseline disease severity (mild, moderate, severe); Test type: Superiority or Other; p = 0.29, Regression, Logistic — Treatment sequence effect: p=0.34; baseline disease severity effect: p=0.29; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and baseline disease severity as factors
Statistical Analysis 4: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: distribution phenotype (localised, widespread); Test type: Superiority or Other; p = 0.55, Regression, Logistic — Treatment sequence effect: p=0.33; distribution phenotype (localised, widespread) effect: p=0.55; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and distribution phenotype (localised, widespread) as factors
Statistical Analysis 5: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: plaque size (≤3 mm diameter, >3 mm diameter); Test type: Superiority or Other; p = 0.25, Regression, Logistic — Treatment sequence effect: p=0.32; plaque size (≤3 mm diameter, >3 mm diameter): p=0.25; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and plaque size as factors
Statistical Analysis 6: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: skin thickness phenotype (≤0.75 mm, >0.75 mm); Test type: Superiority or Other; p = 0.41, Regression, Logistic — Treatment sequence effect: p=0.34; skin thickness phenotype (≤0.75 mm, >0.75 mm) effect: p=0.41; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and skin thickness phenotype as factors
Statistical Analysis 7: Comparison: Foam - Gel vs Gel - Foam; The statistical significance of each of the 7 baseline characteristics was tested in a 2-factor logistic regression model with treatment sequence and each baseline characteristic as factors. Baseline factor: onset phenotype (≤40 years of age, >40 years of age); Test type: Superiority or Other; p = 0.20, Regression, Logistic — Treatment sequence effect: p=0.30; onset phenotype (≤40 years of age, >40 years of age) effect: p=0.20; threshold for statistical significance: p<0.05; 2-factor logistic regression model with treatment sequence and onset phenotype (≤40 years of age, >40 years of age) as factors

2. Other Pre Specified Outcome: Within Subject Difference in Response to Topical Product Usability Questionnaire (TPUQ) Items Between Trial Treatments
Description: Each response category (item 1 to 25) was assigned a numeric score (-2=strongly disagree, -1=slightly disagree, 0=neither agree nor disagree, 1=slightly agree, 2=strongly agree). For item 26, the assigned score were from -2=very dissatisfied to 2=very satisfied.
  Summary scores were calculated by summing numeric scores for items under each domain, i.e., application (items 1-9; score range -18 to +18), formulation (items 10-18; score range -18 to +18), container (items 19-22; score range -8 to +8), and satisfaction (items 23-25; score range -6 to +6). Positive scores indicate agreement with domains' items.
  A total TPUQ summary score (item 1-25; score range -50 to +50) was also calculated. The summary scores were analysed in the same way as the individual questions. The higher score signifies higher preference in that domain.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LEO 90100 Areosol Foam: Subject assessments of LEO 90100 aerosol foam. This column shows LEO 90100 foam assessments from the foam-gel group as well as the gel-foam group.
- Daivobet® Gel: Subject assessments of Daivobet® gel. This column shows Daivobet® gel assessments from the foam-gel group as well as the gel-foam group.
Arm/Group | LEO 90100 Areosol Foam | Daivobet® Gel
Number analyzed (Participants) | 212 | 212
units on a scale
  1. Ease of application | 1.1 (1.2) | 1.5 (0.9)
  2. Ease of application on psoriasis lesions only | 0.9 (1.3) | 1.4 (0.9)
  3. Ease of spreading | 1.5 (0.8) | 1.7 (0.7)
  4. Lack of mess when applying | 0.8 (1.2) | 1.0 (1.2)
  5. Good for use on smaller areas | 1.0 (1.2) | 1.4 (0.9)
  6. Good for use on larger areas | 1.4 (0.9) | 1.5 (0.8)
  7. Quick to apply | 1.4 (0.8) | 1.4 (0.9)
  8. Total time spent acceptable | 1.5 (0.7) | 1.5 (0.8)
  9. Easily incorporated into daily routine | 1.4 (0.9) | 1.5 (0.9)
  Total application score (summary score item 1-9) | 11.1 (6.9) | 12.8 (6.1)
  10. Quickly absorbed | 0.7 (1.3) | 0.7 (1.3)
  11. Dried quickly | 0.5 (1.3) | 0.5 (1.3)
  12. Gave an immediate feeling of relief | 1.0 (1.0) | 0.7 (1.0)
  13. Felt soothing to my skin | 1.2 (1.0) | 1.0 (0.9)
  14. Appealing to touch | 0.9 (1.1) | 0.9 (1.1)
  15. Felt moisturising to my skin | 1.1 (1.0) | 1.2 (0.9)
  16. Not greasy | 0.0 (1.5) | 0.3 (1.4)
  17. Odourless | 1.3 (1.0) | 1.6 (0.7)
  18. Lack of staining of clothes/bed linen | 1.0 (1.3) | 1.0 (1.3)
  Total formulation score (summary score item 10-18) | 7.7 (7.2) | 8.0 (7.4)
  19. Easy to get medication out of container | 1.1 (1.2) | 1.3 (1.0)
  20. Easy to use container | 1.1 (1.2) | 1.4 (0.9)
  21. Easy to keep container clean | 1.2 (1.1) | 1.4 (1.0)
  22. Accurately dispense wanted amount | 0.9 (1.2) | 1.5 (0.9)
  Total container score (summary score item 19-22) | 4.3 (3.8) | 5.6 (3.3)
  23. Confidence in using the product | 1.2 (1.1) | 1.2 (1.0)
  24. Would regularly use the product | 1.3 (1.2) | 1.3 (1.0)
  25. Would recommend the product | 1.2 (1.1) | 1.1 (1.1)
  Total satisfaction score(summary score item 23-25) | 3.6 (3.2) | 3.7 (2.9)
  Total TPUQ score (summary score item 1-25) | 26.8 (17.8) | 29.9 (16.9)
  26. Overall satisfaction score | 1.1 (1.0) | 1.2 (1.0)
Statistical Analysis 1: Comparison: LEO 90100 Areosol Foam vs Daivobet® Gel; Subjects in the analysis are 212 - full analysis set. All subjects received both study treatments. Total TPUQ score (summary score item 1-25) superiority comparison gel versus foam; Test type: Superiority or Other; p = 0.007, Wilcoxon Rank Sum Test — The total TPUQ score for the gel and the foam (mean score 29.9 vs. mean score 26.8; p=0.007). Threshold for statistical significance: p<0.05; Wilcoxon rank sum test comparing the period difference (within subject difference between study treatments) between both treatment sequences

3. Other Pre Specified Outcome: Within Subject Difference in Response to TPUQ Between the Last Topical Anti-psoriatic Treatment and Each of the 2 Trial Treatments
Description: The TPUQ tool was used to evaluate the subject's latest topical treatment at Baseline (used within 3 months prior to baseline). TPUQ assessments of trial treatments at Week 1 and Week 2.
  Each response category (item 1 to 25) was assigned a numeric score from-2=strongly disagree to 2=strongly agree. For item 26 the assigned scores were from -2=very dissatisfied to 2=very satisfied.
  Summary scores were calculated by summing numeric scores for items under each domain, i.e., application (items 1-9; score range -18 to +18), formulation (items 10-18; score range -18 to +18), container (items 19-22; score range -8 to +8), and satisfaction (items 23-25; score range -6 to +6).
  For each subject and each item, the latest topical treatment score was compared with each study treatment by calculating the difference between the scores, i.e., by subtracting the latest topical treatment score from each study medication score. The higher score signifies higher preference in that domain.
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Latest Topical Treatment: Subjects who had used topical treatment to treat their psoriasis within 3 months prior to baseline. Assessments of last topical treatment (TPUQ tool) at baseline.
- LEO 90100 Aerosol Foam: Subjects who had used topical treatment to treat their psoriasis within 3 months prior to Baseline.
  Subject assessments of LEO 90100 aerosol foam. This column shows LEO 90100 aerosol foam assessments from the foam-gel group as well as the gel-foam group.
- Daivobet® Gel: Subjects who had used topical treatment to treat their psoriasis within 3 months prior to baseline.
  Subject assessments of Daivobet® gel. This column shows Daivobet® gel assessments from the foam-gel group as well as the gel-foam group.
Arm/Group | Latest Topical Treatment | LEO 90100 Aerosol Foam | Daivobet® Gel
Number analyzed (Participants) | 118 | 118 | 118
units on a scale
  Total application score (sum score items 1-9) | 9.9 (6.7) | 11.5 (6.7) | 12.5 (6.7)
  Total formulation score (sum score items 10-18) | 2.8 (7.5) | 8.3 (7.2) | 7.5 (8.0)
  Total container score (sum score items 19-22) | 4.6 (3.7) | 4.6 (3.4) | 5.5 (3.4)
  Total satisfaction score (sum score items 23-25) | 2.0 (3.0) | 4.0 (3.0) | 3.4 (3.2)
  Total TPUQ score (items 1-25) | 19.4 (16.9) | 28.4 (17.1) | 29.0 (18.6)
  26. Overall satisfaction score | 0.3 (1.1) | 1.2 (1.0) | 1.1 (1.1)
Statistical Analysis 1: Comparison: Latest Topical Treatment vs LEO 90100 Aerosol Foam; Subjects in the analysis are 118. All subjects received both study treatments. Statistical analysis for total TPUQ score (summary score item 1-25): superiority comparison foam versus latest topical treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test; Wilcoxon signed rank test comparing within subject difference to latest topical treatment
Statistical Analysis 2: Comparison: Latest Topical Treatment vs Daivobet® Gel; Subjects in the analysis are 118. All subjects received both study treatments. Statistical analysis for total TPUQ score (summary score item 1-25): superiority comparison gel versus latest topical treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test; Wilcoxon signed rank test comparing within subject difference to latest topical treatment

4. Other Pre Specified Outcome: Responses to Comparison to Last Topical Treatment Questionnaire (CLTT) for Each of the Two Trial Treatments (Foam or Gel)
Description: Subjects in both arms (foam-gel; gel-foam) indicated whether they preferred latest topical treatment, LEO 90100 aerosol foam, Daivobet® gel, or did not have any preference.
  The subjects compared the trial treatment used the previous week with the latest topical treatment (used within 3 months prior to baseline; CLTT analysis set). Each item was scored with either 'prefer latest treatment', 'no preference', or 'prefer trial medication (foam or gel)'. A subject could prefer both study treatments over the latest topical treatment. The percentage is given for the number of subjects preferring foam and number of subjects preferring gel.
Time Frame: At Week 1 and Week 2
Population: CLTT analysis set was defined by including all randomised subjects who had used topical anti-psoriatic medication on the treatment area (trunk and/or limbs) within 3 months prior to Baseline.
Measure: Number; unit: percentage of subjects
Groups:
- All Subjects Foam: Subject assessments of LEO 90100 aerosol foam compared to latest topical treatment (CLTT analysis set).
- All Subjects Gel: Subject assessments of Daivobet® gel compared to latest topical treatment (CLTT analysis set).
Arm/Group | All Subjects Foam | All Subjects Gel
Number analyzed (Participants) | 118 | 118
percentage of subjects | 76.5 | 70.2

5. Other Pre Specified Outcome: Within Subject Difference in Response to Vehicle Preference Measure (VPM) Items Between Trial Treatments
Description: The VPM questionnaire was analysed the same way as the TPUQ. Numeric scores were calculated by assigning the following values to each response category: -3 = Extremely unappealing, -2 = Moderately unappealing, -1 = Slightly unappealing, 0 = Neutral, 1 = Slightly appealing, 2 = Moderately appealing, 3 = Extremely appealing. A summary score was defined as the sum of all questions and could range from -21 to 21.
Time Frame: At Week 1 and Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 90100 Areosol Foam | Daivobet® Gel
Number analyzed (Participants) | 212 | 212
units on a scale
  Ease of application | 1.5 (1.7) | 1.9 (1.4)
  Time it takes to apply | 1.9 (1.4) | 2.0 (1.4)
  How well it is absorbed | 1.4 (1.6) | 1.4 (1.6)
  How it feels to touch | 1.4 (1.6) | 1.6 (1.4)
  How it smells | 1.6 (1.5) | 1.9 (1.3)
  How it feels on the skin | 1.8 (1.5) | 1.8 (1.4)
  How much it stains | 1.4 (1.5) | 1.3 (1.6)
  Total VPM score (summary score) | 11.1 (7.8) | 12.0 (7.8)

6. Other Pre Specified Outcome: Reasons for Overall Preference as Assessed by Subject's Preference Assessment (SPA) at Week 2
Description: Comparison of contribution of each product attribute in the stated preference between trial treatments (foam and gel)
Time Frame: Baseline to Week 2
Population: In total 103 preferred foam and 105 preferred gel. 4 subjects ...
Measure: Number; unit: percentage of subjects
Groups:
- Prefer Foam - Very Important Factor; Prefer Foam - Fairly Important Factor; Prefer Foam - Not Very Important Factor; Prefer Foam - Not at All Important Factor: Subjects who prefer foam
- Prefer Gel - Very Important Factor; Prefer Gel - Fairly Important Factor; Prefer Gel - Not Very Important Factor; Prefer Gel - Not at All Important Factor: Subjects who prefer gel
Arm/Group | Prefer Foam - Very Important Factor | Prefer Foam - Fairly Important Factor | Prefer Foam - Not Very Important Factor | Prefer Foam - Not at All Important Factor | Prefer Gel - Very Important Factor | Prefer Gel - Fairly Important Factor | Prefer Gel - Not Very Important Factor | Prefer Gel - Not at All Important Factor
Number analyzed (Participants) | 103 | 103 | 103 | 103 | 105 | 105 | 105 | 105
percentage of subjects
  The medication was easy to apply | 51.5 | 30.1 | 12.6 | 5.8 | 54.3 | 37.1 | 4.8 | 3.8
  Easy application on psoriasis lesions only | 48.5 | 31.1 | 14.6 | 5.8 | 61.0 | 30.5 | 4.8 | 3.8
  Easy to spread | 65.0 | 24.3 | 4.9 | 5.8 | 52.4 | 41.0 | 2.9 | 3.8
  Applying the medication was not messy | 47.6 | 34.0 | 15.5 | 2.9 | 45.7 | 44.8 | 4.8 | 4.8
  Overall good for smaller areas | 53.6 | 29.9 | 8.2 | 8.2 | 50.5 | 38.4 | 7.1 | 4.0
  Overall good for larger areas | 61.8 | 25.8 | 5.6 | 6.7 | 44.2 | 44.1 | 10.5 | 3.2
  Treatment was quick to apply | 55.3 | 34.0 | 7.8 | 2.9 | 45.7 | 45.7 | 4.8 | 3.8
  Total time spent on treatment acceptable | 57.3 | 26.2 | 11.7 | 4.9 | 48.6 | 41.9 | 6.7 | 2.9
  Applying treatment easy in daily routine | 61.2 | 24.3 | 10.7 | 3.9 | 56.2 | 36.2 | 3.8 | 3.8
  Treatment quickly absorbed | 51.5 | 32.0 | 11.7 | 4.9 | 50.5 | 39.0 | 9.5 | 1.0
  Treatment dried quickly | 45.6 | 35.0 | 17.5 | 1.9 | 50.5 | 39.0 | 9.5 | 1.0
  Treatment gave immediate feeling of relief | 48.5 | 31.1 | 18.4 | 1.9 | 39.0 | 41.0 | 17.1 | 2.9
  The medication felt soothing to my skin | 50.5 | 36.9 | 8.7 | 3.9 | 46.7 | 39.0 | 12.4 | 1.9
  The medication was appealing to touch | 44.7 | 34.0 | 14.6 | 6.8 | 34.3 | 39.0 | 21.0 | 5.7
  Treatment felt moisturising to my skin | 45.6 | 38.8 | 11.7 | 3.9 | 41.0 | 43.8 | 12.4 | 2.9
  Treatment not too greasy | 48.5 | 30.1 | 17.5 | 3.9 | 43.8 | 38.1 | 15.2 | 2.9
  Treatment was odourless | 46.6 | 26.2 | 18.4 | 8.7 | 38.1 | 41.0 | 16.2 | 4.8
  Absence of staining of clothes/bed linen | 53.4 | 31.1 | 11.7 | 3.9 | 54.3 | 36.2 | 7.6 | 1.9
  Getting treatment out of container | 52.4 | 32.0 | 10.7 | 4.9 | 52.4 | 41.0 | 2.9 | 3.8
  Container easy to use | 55.3 | 31.1 | 10.7 | 2.9 | 57.1 | 36.2 | 4.8 | 1.9
  Ease of keeping clean container | 42.7 | 33.0 | 16.5 | 7.8 | 45.7 | 38.1 | 16.2 | 0.0
  Dispensing the desired amount | 54.4 | 34.0 | 8.7 | 2.9 | 59.0 | 33.3 | 5.7 | 1.9

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: 21 subjects (9.9%) experienced a total of 21 treatment-emergent AEs. No SAEs, severe AEs or AEs leading to withdrawal were observed. 2 subjects had AEs which were assessed as related to study treatment by the investigator: one subject in the foam-gel group experienced folliculitis, and one subject in the gel-foam group experienced dermatitis.
Arm/Group | Foam - Gel | Gel - Foam
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/104
Other Adverse Events (participants affected / at risk) | 13/109 | 8/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foam - Gel (N=109) | Gel - Foam (N=104)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Arthroscopy (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.